CLINICAL TRIAL: NCT04319601
Title: A Single-arm, Multiple Centers, Phase II Study Evaluating Rituximab in Combination With Chidamide and Lenalidomide for Relapsed or Refractory Angioimmunoblastic T-cell Lymphoma (AITL)
Brief Title: Rituximab Combined With Chidamide and Lenalidomide for r/r AITL
Acronym: AITL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhejiang Cancer Hospital (Other)
Responsible Party: Principal Investigator, Yang haiyan, Head of lymphoma oncology, Zhejiang Cancer Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RLC
Record Dates: First submitted 2020-03-10; First posted 2020-03-24 (Actual); Last update posted 2021-03-24 (Actual); Status verified 2020-03

CONDITIONS: Angioimmunoblastic T-cell Lymphoma; Chemotherapy Effect; Chemotherapeutic Toxicity
MeSH Terms: conditions — Immunoblastic Lymphadenopathy | interventions — Rituximab; N-(2-amino-5-fluorobenzyl)-4-(N-(pyridine-3-acrylyl)aminomethyl)benzamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- rituximab combined with chidamde and lenalidomide (Experimental): rituximab and chidamide, lenalidomide
  Interventions: Drug: Rituximab

INTERVENTIONS:
Drug: Rituximab — a new chemotherapy regimen
  Other Names: chidamide; lenalidomde

SUMMARY:
This study is designed to explore the effeicency and toxicities of rituximab combined with chidamide and lenalidomide in patients with relapsed or refractory AITL.

DETAILED DESCRIPTION:
This study is designed to explore the effeicency and toxicities of rituximab combined with chidamide and lenalidomide in patients with relapsed or refractory AITL. The primary end point is PFS, and second end point is OS, ORR and toxicities according to CTCAE 5.0.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must voluntarily participate in this study and sign an informed consent.
2. 18-70 years old.
3. ECOG 0-2.
4. Life expectancy ≥12 weeks.
5. Histopathology diagnosis of AITL.
6. A measurable lesion (lymphoma nodule, lymph node mass or other lymphoma lesions as defined in lugano 2014) that can be measured in both diameters on the CT scan, including the longest diameter and the shortest diameter perpendicular to the longest diameter.In addition, the longest diameter of lymph nodes should be greater than 1.5cm, and the longest diameter of external lymph node lesions should be greater than 1.0cm.
7. The patient has received at least one line of systemic chemotherapy and currently has disease progression or treatment failure, or the patient refuses or cannot tolerate intravenous chemotherapy.
8. Adequate bone marrow hematopoietic function reserve and viscera function, as follows:

Liver function: ALT, AST≤2.5 times the normal upper limit, if there is liver metastasis, ≤5 times the normal upper limit;Total bilirubin, direct bilirubin ≤1.5 times the normal upper limit.

Bone marrow function (growth factor should not be used within 7 days before the first medication) : WBC ≥2.0*109/l;The ANC acuity 1.0 * 109 / l;PLT 50 * 109 / l or higher;Hb 8 g/dl or higher.

Renal function: creatinine ≤1.5 times the normal upper limit or creatinine clearance ≥30ml/min.

Cardiac function: LVEF≥50%. Lung function: resting and oxygen saturation ≥95% without oxygen inhalation. Coagulation function: international standardized ratio (INR) ≤1.5×ULN and activated partial thromboplastin time (aPTT) ≤1.5×ULN, unless the patient is receiving anticoagulation therapy and the coagulation parameters (prothrombin time [PT/INR] and aPTT) at the time of screening are within the expected range of anticoagulant treatment.Patients whose prolongation of PT or elevation of INR resulted from the use of clotting factor inhibitors were eligible for inclusion by the investigator.

Exclusion Criteria:

1. Prior to the first use of the drug in this study, there was an unrelieved drug toxicity greater than CTCAE1 (except for the adverse reactions, such as hair loss, that the investigator assessed did not affect the use of the drug in this study).
2. Presence of active infection, including but not limited to: known active/latent tuberculosis, herpes zoster, pneumonia.

3, Known human immunodeficiency virus (HIV) infection, or reflect the activity of hepatitis b virus (HBV) or hepatitis c virus (HCV) infection of serological status: a. the hepatitis b surface antigen (HBsAg) positive, HBcAb positive, HBsAg positive patients should be detected HBV - DNA, if not more than 1000 iu/ml and agreed to accept patients treated against HBV virus can enter the group.B. patients with positive HCV antibody are admitted if HCV RNA (<15 IU/mL) is not detected.

4. Patients with heart failure of grade 3 or 4 according to the New York society of cardiology (NYHA) functional classification, unstable angina, severe poorly controlled ventricular arrhythmia, electrocardiogram showing acute ischemia or myocardial infarction 6 months prior to screening.Or other cardiac dysfunction assessed by the investigator as not resistant to chemotherapy.

5. Support the treatment of refractory nausea, vomiting, chronic gastrointestinal diseases, capsule dysphagia, or previous surgical resection of the intestinal segment may affect the full absorption of drugs.

6. The investigator's judgment or other evidence indicates that the patient has serious or poorly controlled systemic diseases, including poorly controlled hypertension and an active bleeding constitution.At present, patients with thrombotic diseases such as pulmonary embolism and deep vein thrombosis are also not suitable to participate in this study.

7. Nursing or pregnant women. 8. The researcher judged that the patient had other factors that might affect the compliance of the plan.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2020-03-13 (Actual); Primary Completion 2022-03-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
PFS | From enrollment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 32 months
  progression free survival

SECONDARY OUTCOMES:
ORR | From enrollment until date of completion of chemotherapy, assessed up to 9 months
  overall response rate
toxicities | from enrollment to 30 days after completion of chemotherapy, assessed up to 9 months
  Number of participants with treatment-related adverse events as assessed by CTCAE v5.0

CONTACTS AND LOCATIONS:
Overall Officials: Ming Chen, PhD, Study Chair — Zhejiang Cancer Hospital
Locations (1):
- Zhejiang Cancer Hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No